CLINICAL TRIAL: NCT01954173
Title: Phase II Study of Adjuvant 3D-Conformal Radiotherapy in High Risk Bladder Cancer
Brief Title: Adjuvant Radiation for High Risk Bladder Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Joseph W Shelton MD, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00059097; NCI-2013-01381 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RAD2271-12 (Other: Emory University)
Record Dates: First submitted 2013-08-19; First posted 2013-10-01 (Estimated); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Bladder Cancer; Squamous Cell Carcinoma of the Bladder; Stage III Bladder Cancer; Stage IV Bladder Cancer; Transitional Cell Carcinoma of the Bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 3D conformal radiation therapy (Experimental): Within 24 weeks of surgical resection, patients undergo conformal radiation therapy once daily 5 days per week for 28 fractions. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: 3D conformal radiation therapy

INTERVENTIONS:
Radiation: 3D conformal radiation therapy — Undergo conformal radiation therapy
  Other Names: 3D-CRT; IMRT; Intensity Modulated Radiotherapy

SUMMARY:
This phase II trial studies how well modern, conformal radiation therapy after surgery works in treating patients with high-risk bladder cancer. Specialized radiation therapy that delivers a high dose of radiation directly to the tumor may kill more tumor cells and cause less damage to normal tissue.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine the feasibility of adjuvant radiation in the management of high-risk disease.

SECONDARY OBJECTIVES:

I. Prospectively evaluate patterns of failure in high-risk bladder cancer patients after cystectomy and aggressive adjuvant therapy.

II. Define surgical and histopathologic parameters predictive of local and distant outcomes (e.g. grade, lymphovascular space invasion [LVSI], extent of resection/lymph node dissection [LND]).

III. Assess quality of life (QoL) outcomes after this treatment using a standardized questionnaires (Functional Assessment of Cancer Therapy-General [FACT-G], FACT-Bladder Cancer [BL], Expanded Prostate Cancer Index Composite [EPIC] Bowel and Urinary).

OUTLINE:

Within 24 weeks of surgical resection, patients undergo 3D conformal radiation therapy once daily 5 days per week for 28 fractions. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4 weeks, every 3 months for 2 years, every 6 months for 3-5 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Pathologic diagnosis of urothelial or squamous cell carcinoma of the bladder
* Patients must have undergone cystectomy (total cystectomy, radical cystectomy +/- pelvic lymph node dissection) with no evidence of macroscopic residual disease
* Eastern Cooperative Oncology Group (ECOG)/Zubrod performance status of 0-2
* Patients treated with simple cystectomy with macroscopically negative margins are eligible for this study
* Clinical T-stage (prior to systemic therapy, if applicable) ≥ T3a and/or positive lymph nodes by transurethral resection of bladder tumor (TURBT)/magnetic resonance imaging (MRI)/computed tomography (CT)/positron emission tomography (PET)-CT or pathologic T-stage ≥ T3a and/or positive lymph nodes

Exclusion Criteria:

* Patients with metastatic disease outside of the pelvis
* Prior invasive malignancy (except non-melanomatous skin cancer) unless disease free for a minimum of 3 years
* Prior radiation therapy to the pelvis
* Patients with active inflammatory bowel disease
* Severe acute co-morbidity, defined as follows:

  * Unstable angina and/or congestive heart failure requiring hospitalization in the last 3 months
  * Transmural myocardial infarction within the last 6 months
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
  * Acquired immune deficiency syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; note, however, that human immunodeficiency virus (HIV) testing is not required for entry into this protocol; the need to exclude patients with AIDS from this protocol is necessary because the treatment involved in this protocol may be significantly immunosuppressive; protocol-specific requirements may also exclude immunocompromised patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-07-22 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal (GI) late effects, assessed using Radiation Therapy Oncology Group (RTOG) Late Effects in Normal Tissues (LENT)/Subjective, Objective, Management and Analytic (SOMA) scales | 3 months to 10 yrs
  For purposes of this study, "bowel adverse events" are defined as the following: diarrhea, enteritis, fistula, ileus, incontinence, obstruction, perforation, proctitis, and stricture/stenosis (including anastomotic) as graded buy Common Terminology for Adverse Events (CTCAE) version 4.0.

SECONDARY OUTCOMES:
Acute adverse events greater than grade 2, graded by CTCAE version 4.0 | Up to 90 days
Loco-regional failure, considered any failure in the treatment field of the pelvis | Up to 5 years
  The cumulative incidence approach will be used to estimate the failure rate for local-regional and distant failures.
Rate of distant metastases | Up to 5 years
  Nodal disease beyond the common iliac will be considered distant failure. The cumulative incidence approach will be used to estimate the failure rate for distant failure.
Rate of disease-free survival | Up to 5 years
  Any tumor recurrence, development of distant metastases or death is considered a failure. The Kaplan-Meier method will be used to estimate the disease-free survival rate.
Overall survival rate | Up to 5 years
  Death from any cause is considered a failure. The Kaplan-Meier method will be used to estimate the overall survival.
Quality of life, assessed using FACT-BL | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joseph W Shelton, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States